CLINICAL TRIAL: NCT06018740
Title: A Single Group Clinical Trial to Examine the Effects of a Daily Supplement on Common Symptoms of Perimenopause and Menopause
Brief Title: A Study to Examine the Effects of a Daily Supplement on Common Symptoms of Perimenopause and Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hologram Sciences (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20356
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Menopause; Perimenopause

STUDY DESIGN:
Intervention Model Description: Single group clinical trial.
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily Balance Gummy (Experimental): One Daily Balance Gummy should be taken with the last meal of the day.
  Interventions: Dietary Supplement: Daily Balance Gummy

INTERVENTIONS:
Dietary Supplement: Daily Balance Gummy — Phenology Daily Balance Gummies 30 ct. Yuzu Tangerine Flavor. Product contains Vitamin D2, Vitamin K2, Vitamin B6, Vitamin B12, Biotin, Genistein, Saffron Extract, Organic Tapioca Syrup, Organic Cane Sugar, Water, Pectin, Citric Acid, Natural Flavors.

SUMMARY:
Symptoms of perimenopause and menopause can significantly affect overall quality of life. It is hypothesized that daily supplements can reduce the severity of these symptoms. This 12-week clinical trial will examine the effects of Hologram Sciences' Daily Balance Gummy Supplements on symptoms including hot flashes, night sweats, mood swings, anxiety, fatigue, and brain fog. Participants will take the product daily and complete study-specific questionnaires at Baseline, Week 4, Week 8, and Week 12. Upon conclusion of Week 12, participants will be asked to count how many gummies remain in their jar.

ELIGIBILITY:
Inclusion Criteria:

Women aged 40-65 years old Must be experiencing at least two symptoms of menopause, such as sleep disturbances, mood changes, fatigue and lack of energy, changes in sexual function, urinary changes, irregular or absent periods, or vaginal changes Must experience hot flashes and/or night sweats at least 5 times per day Can be either natural or surgical menopause (or perimenopause) Willing to adhere to the study protocol for the duration of the study

Willing to consult with their physician prior to starting the trial if taking any of the following medications:

Levothyroxine Liothyronine Calcipotriene (Dovonex) Digoxin (Lanoxin) Diltiazem (Cardizem) Verapamil (Calan, others) Thiazide diuretics Atorvastatin (Lipitor) Warfarin - Might increase the amount of time it takes for blood clotting. Minosalicylic acid (Paser) Colchicine (Colcrys, Mitigare, Gloperba) Metformin (Glumetza, Fortamet, others) Proton pump inhibitors (omeprazole (Prilosec), lansoprazole (Prevacid) or other stomach acid-reducing drugs) Phenytoin (Dilantin) Antihypertensive drugs Phenobarbital (Luminal) Amiodarone (Cordarone) Levodopa

Exclusion Criteria:

Not experiencing hot flashes and/or night sweats at least 5 times per day Has taken herbal supplements or multivitamins within the last 1 month Current use of conventional hormone replacement therapies, or plan to start during the study duration Current use of hormonal birth control, or plan to start during the study duration Known allergies to any product ingredients including the purified isoflavone genistein History of uterine fibroids, endometriosis, polycystic ovarian syndrome, or history of abnormal pap smear Anyone with any known severe allergies requiring the use of an epi-pen Unwilling to adhere to the study protocol Anyone living with uncontrolled or chronic health disorders, including oncological or psychiatric disorders No planned invasive medical procedures for the duration of the study Pregnant or breastfeeding

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Changes in score on the Menopause Rating Scale (MRS). [Baseline to Week 12] | 12 weeks
  The Menopause Rating Scale (MRS) is a commonly used assessment tool in medical and research settings to evaluate the severity and impact of menopausal symptoms on women's lives. 5 point Likert scale, with the following points relating to menopausal symptoms: 0 - None (absent)
  1. - Mild (light)
  2. - Moderate (medium)
  3. - Severe (heavy)
  4. - Very severe (very heavy)
Change in hot flashes. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in hot flashes. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('Extremely often') and 5 representing the most beneficial response (i.e., "never").
Change in night sweats. [Baseline to 12 Weeks] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in night sweats. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('severe') and 5 represents the most beneficial response (i.e., "not noticeable").
Change in brain fog. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in brain fog. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('severe') and 5 represents the most beneficial response (i.e., "not noticeable").
Change in mood swings. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in mood swings. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('severe') and 5 represents the most beneficial response (i.e., "not noticeable").
Change in sleep disturbances. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in sleep disturbances. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('severe') and 5 represents the most beneficial response (i.e., "not noticeable").
Change in fatigue. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of changes in fatigue. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('severe') and 5 represents the most beneficial response (i.e., "not noticeable").

SECONDARY OUTCOMES:
Changes in participant-reported quality of life. [Baseline to Week 12] | 12 weeks
  Survey-based assessment (0-5 point scale) of quality of life. The survey has been designed specifically for use in this study and includes study-specific questions. Data will be collected using a textual 5-point Likert scale for each question, such as "Not noticeable" to "severe." A score of 0 represents the least favorable/worse outcome ('Very Poor') and 5 represents the most beneficial response (i.e., "Excellent").

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided